CLINICAL TRIAL: NCT00577226
Title: Use of the Shilla Growth Permitting Spinal Instrumentation System/Technique for the Treatment of Scoliosis in the Immature Spine
Brief Title: Shilla Growth Permitting Spinal Instrumentation System for Treatment of Scoliosis in the Immature Spine
Status: Terminated | Type: Observational
Why Stopped: IRB has requested additional information regarding IDE
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 32975
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Scoliosis
Keywords: scoliosis, immature spine
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 Shilla Technique: The patients whose data is observed are those who have undergone the shilla surgical technique.

SUMMARY:
The objective of this study is to retrospectively and prospectively review patients who have undergone this technique looking at age of the patient, magnitude of the curve preoperatively, postoperatively and over time, diagnosis, pulmonary function, surgical procedures, complications, and spinal growth.

The hypothesis is that Shilla growth permitting spinal instrumentation coupled with a surgical technique of aggressive correction of the apex of the scoliotic curve wil allow for natural growth of the spine in a guided fashion with a limited number of future surgeries required.

DETAILED DESCRIPTION:
Traditional "growing rod" constructs of spinal instrumentation to treat severe scoliosis in young children require a return to the operating room every six to nine months until skeletal maturity. The Shilla system allows for more spinal growth with fewer surgical procedures necessary for lengthenings. This is a major advantage over existing growth permitting systems and allows surgery to be performed at younger ages with better deformity correction without concerns of repeated surgeries.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 1 yr and 10 yrs
* have severe, progressive scoliosis unresponsive to bracing
* have severe, progressive scoliosis who cannot tolerate bracing

Exclusion Criteria:

* none

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients whose data is observed are those who have undergone the shilla surgical technique.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patients treated with Shilla procedure will undergo fewer surgeries than patients treated with traditional growing rod constructs. | 5 yrs

SECONDARY OUTCOMES:
Patients will have continued spinal growth | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. McCarthy, M.D., Principal Investigator — University of Arkansas for Medical Sciences/Arkansas Childrens Hospital
Locations (1):
- Arkansas Childrens Hospital, Little Rock, Arkansas, United States